CLINICAL TRIAL: NCT01063699
Title: Prospective Trial on Survival With Own Liver After Conventional Versus Laparoscopic Kasai for Biliary Atresia
Brief Title: Survival With Own Liver of Conventional Versus Laparoscopic Kasai for Biliary Atresia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Benno M Ure, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBAR 9260
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-12

CONDITIONS: Biliary Atresia
Keywords: biliary atresia - laparoscopy - kasai - portoenterostomy
MeSH Terms: conditions — Biliary Atresia | interventions — Portoenterostomy, Hepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lap Kasai (Experimental): Patients in this arm had their necessary Kasai procedure in a laparoscopic way.
  Interventions: Procedure: Laparoscopic Kasai operation

INTERVENTIONS:
Procedure: Laparoscopic Kasai operation — the Kasai procedure (hepatoportoenterostomy) is performed laparoscopically, thus not in open surgery.
  Other Names: hepatoportoenterostomy; coelioscopie

SUMMARY:
This study evaluated laparoscopic (videosurgery) versus conventional (open surgery) Kasai portoenterostomy (anastomosis of small intestine to the liver hilus) in children with biliary atresia. The study was stopped due to lower survival with native liver 6 months after the laparoscopic operation. Follow-up after 24 months confirmed superior results after conventional operation.

DETAILED DESCRIPTION:
Objective:

A prospective observational study to compare survival with own liver in laparoscopic versus conventional Kasai portoenterostomy in patients with biliary atresia.

Summary Background Data:

Available studies on laparoscopic versus conventional Kasai portoenterostomy focus on short-term results, include limited numbers of patients and have design limitations.

Methods:

A consecutive series of patients underwent laparoscopic Kasai procedure from 2006 to 2007. Conventionally operated control patients consisted of a consecutive series of infants with biliary atresia operated from August 2003 to 2006. All data were ascertained prospectively using the European Biliary Atresia Registry / EBAR registration forms. Primary outcome measure was survival with own liver 6 months after Kasai without being listed for liver transplantation. An interim analysis was planned after data became available for the first 12 patients who underwent laparoscopic Kasai procedure. In case of a significantly different interim outcome the follow-up period should be extended to 24 months until a final decision should be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Biliary atresia

Exclusion Criteria:

* < 3000 grs. body weight
* Syndromatic form of biliary atresia
* Significant comorbidity i.e. cardiac
* Contraindication to laparoscopy

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2003-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Survival with own liver at 6 months after the Kasai operation without beeing listed for liver transplantation | one year

SECONDARY OUTCOMES:
Jaundice free survival confirmed by serum bilirubin < 20 umol/l | 6 months
Feasibility of laparoscopic Kasai with regard to conversions and revisions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Petersen, Prof., Study Director — MHH pediatric surgery
Locations (1):
- Hannover Medical School Pediatric Surgery Dpmt., Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] FUJINO M, KASAI K, KOSEKI A. The effects of temperature on actomyosin adenosinetriphosphatase activity and super-precipitation. Jpn J Physiol. 1959 Jun 25;9(2):228-38. doi: 10.2170/jjphysiol.9.228. No abstract available. PMID 13672695
- [Background] Okazaki T, Miyano G, Yamataka A, Kobayashi H, Koga H, Lane GJ, Miyano T. Diagnostic laparoscopy-assisted cholangiography in infants with prolonged jaundice. Pediatr Surg Int. 2006 Feb;22(2):140-3. doi: 10.1007/s00383-005-1609-0. Epub 2005 Dec 8. PMID 16341535
- [Derived] Ure BM, Kuebler JF, Schukfeh N, Engelmann C, Dingemann J, Petersen C. Survival with the native liver after laparoscopic versus conventional kasai portoenterostomy in infants with biliary atresia: a prospective trial. Ann Surg. 2011 Apr;253(4):826-30. doi: 10.1097/SLA.0b013e318211d7d8. PMID 21475026